CLINICAL TRIAL: NCT06080581
Title: Mitochondrial Derangements Driving Muscle Insulin Resistance in Humans
Brief Title: Mitochondrial Dysfunctions Driving Insulin Resistance
Acronym: MITO-DYS-IR
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Matteo Fiorenza, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: MITO-DYS-IR
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Mitochondrial Myopathies; Mitochondrial Diseases; Mitochondrial Disorders
Keywords: Mitochondrial disease; Muscle metabolism; Insulin resistance
MeSH Terms: conditions — Mitochondrial Myopathies; Mitochondrial Diseases; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, muscle tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mitochondrial myopathy: Individuals with pathogenic mtDNA mutations
- Control: Individuals without mtDNA mutations

SUMMARY:
The overarching aim of this observational study is to characterize muscle mitochondrial defects in individuals harboring pathogenic mitochondrial DNA (mtDNA) mutations associated with an insulin-resistant phenotype.

In a case-control design, individuals with pathogenic mtDNA mutations will be compared to controls matched for sex, age, and physical activity level. Participants will attend a screening visit and two experimental trials including:

* An oral glucose tolerance test
* A hyperinsulinemic-euglycemic clamp combined with measurements of femoral artery blood flow and arteriovenous difference of glucose
* Muscle biopsy samples

DETAILED DESCRIPTION:
Background: Peripheral insulin resistance is a major risk factor for metabolic diseases such as type 2 diabetes. Skeletal muscle accounts for the majority of insulin-stimulated glucose disposal, hence restoring insulin action in skeletal muscle is key in the prevention of type 2 diabetes. Mitochondrial dysfunction is implicated in the etiology of muscle insulin resistance. Also, as mitochondrial function is determined by its proteome quantity and quality, alterations in the muscle mitochondrial proteome may play a critical role in the pathophysiology of insulin resistance. However, insulin resistance is multifactorial in nature and whether mitochondrial derangements are a cause or a consequence of impaired insulin action is unclear. In recent years, the study of humans with genetic mutations has shown enormous potential to establish the mechanistic link between two physiological variables; indeed, if the mutation has a functional impact on one of those variables, then the direction of causality can be readily ascribed. Mitochondrial myopathies are genetic disorders of the mitochondrial respiratory chain affecting predominantly skeletal muscle. Mitochondrial myopathies are caused by pathogenic mutations in either nuclear or mitochondrial DNA (mtDNA), which ultimately lead to mitochondrial dysfunction. Although the prevalence of mtDNA mutations is just 1 in 5,000, the study of patients with mtDNA defects has the potential to provide unique information on the pathogenic role of mitochondrial derangements that is disproportionate to the rarity of affected individuals. The m.3243A>G mutation in the MT-TL1 gene encoding the mitochondrial leucyl-tRNA 1 gene is the most common mutation leading to mitochondrial myopathy in humans. The m.3243A>G mutation is associated with impaired glucose tolerance and insulin resistance in skeletal muscle. Most importantly, insulin resistance precedes impairments of β-cell function in carriers of the m.3243A>G mutation, making these patients an ideal human model to study the causative nexus between muscle mitochondrial dysfunction and insulin resistance. Thus, a comprehensive characterization of mitochondrial functional defects and the associated proteome alterations in patients harboring a mtDNA mutation associated with an insulin-resistant phenotype may elucidate the causal nexus between mitochondrial derangements and insulin resistance. Also, as mitochondrial dysfunction exhibits many faces (e.g. reduced oxygen consumption rate, impaired ATP synthesis, overproduction of reactive oxygen species, altered membrane potential), such an approach may clarify which features of mitochondrial dysfunction play a prominent role in the pathogenesis of insulin resistance.

Objective: To characterize muscle mitochondrial defects in individuals harboring pathogenic mitochondrial DNA (mtDNA) mutations associated with an insulin-resistant phenotype.

Study design: Case-control study in individuals with pathogenic mtDNA mutations (n=15) and healthy controls (n=15) matched for sex, age, and physical activity level.

Endpoint: Differences between individuals with pathogenic mtDNA mutations and controls.

ELIGIBILITY:
Eligibility criteria for individuals with pathogenic mtDNA mutations

Inclusion criteria:

* Known m.3243A>G mutation in the MT-TL1 gene encoding the mitochondrial leucyl-tRNA 1 gene
* Other known mtDNA point mutations

Exclusion criteria:

* Use of antiarrhythmic medications or other medications which, in the opinion of the investigators, have the potential to affect outcome measures.
* Diagnosed severe heart disease, dysregulated thyroid gland conditions, or other dysregulated endocrinopathies, or other conditions which, in the opinion of the investigators, have the potential to affect outcome measures.
* Pregnancy

Eligibility criteria for controls

Exclusion criteria:

* Current and regular use of antidiabetic medications or other medications which, in the opinion of the investigators, have the potential to affect outcome measures.
* Diagnosed heart disease, symptomatic asthma, liver cirrhosis or -failure, chronic kidney disease, dysregulated thyroid gland conditions or other dysregulated endocrinopathies, or other conditions which, in the opinion of the investigators, have the potential to affect outcome measures
* Daily use of tobacco products
* Excessive alcohol consumption
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with mitochondrial myopathy due to pathogenic mtDNA mutations are identified and recruited from the Copenhagen Neuromuscular Center or the Department of Clinical Genetics (Rigshospitalet).
  Control volunteers are recruited via recruitment announcements in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle insulin sensitivity | 90-150 minutes after initiation of the hyperinsulinemic euglycemic clamp
  Insulin-stimulated muscle glucose uptake is determined by the hyperinsulinemic-euglycemic clamp method integrated with measurements of femoral artery blood flow and arteriovenous difference of glucose
Whole-body insulin sensitivity | 90-150 minutes after initiation of the hyperinsulinemic euglycemic clamp
  Whole-body insulin sensitivity is determined by the hyperinsulinemic-euglycemic clamp method
Muscle mitochondrial respiration | Baseline
  Mitochondrial O2 flux is measured by high-resolution respirometry in permeabilized fibers from muscle biopsy samples
Muscle mitochondrial reactive oxygen species (ROS) production | Baseline
  Mitochondrial H2O2 emission rates are measured by high-resolution fluorometry in permeabilized fibers from muscle biopsy samples
Muscle mitochondrial proteome | Baseline
  Mitochondrial proteome signatures are determined by mass spectrometry-based proteomics in muscle biopsy samples

SECONDARY OUTCOMES:
Glucose tolerance | 0-180 minutes after ingestion of an oral glucose solution
  Glucose tolerance is determined by the plasma glucose response curve measured during an oral glucose tolerance test
Beta cell function | 0-180 minutes after ingestion of an oral glucose solution
  Beta cell function is determined by measurements of plasma insulin and insulin C-peptide during an oral glucose tolerance test
Muscle mtDNA heteroplasmy | Baseline
  mtDNA mutation load is measured in muscle biopsy samples from the patients with mitochondrial myopathy
Muscle insulin signaling | Before (baseline) and 0-150 minutes after initiation of a hyperinsulinemic-euglycemic clamp
  Insulin-mediated changes in the abundance of (phosphorylated) proteins modulating insulin action are measured by immunoblotting in muscle and fat biopsy samples
Muscle integrated stress response signaling proteins | Baseline
  Abundance of (phosphorylated) proteins modulating the integrated stress response pathway is measured by immunoblotting in muscle biopsy samples.
Muscle integrated stress response genes | Baseline
  mRNA content of genes governing the integrated stress response pathway is measured by Real-Time PCR in muscle biopsy samples.
Muscle release of FGF21 and GDF15 | Before (baseline) and 0-150 minutes after initiation of a hyperinsulinemic-euglycemic clamp
  Skeletal muscle production of FGF21 and GDF15 is determined by measurements of femoral artery blood flow and arteriovenous difference of plasma FGF21 and GDF15

OTHER OUTCOMES:
Body composition | Baseline
  Whole-body fat free mass and fat mass are determined by dual-energy X-ray absorptiometry
Leg muscle mass | Baseline
  Leg muscle mass is determined by dual-energy X-ray absorptiometry
Physical activity level | Baseline
  Physical activity is measured by wrist-worn accelerometers
Self-reported physical activity | Baseline
  Self-reported physical activity is measured by the International Physical Activity Questionnaire - Short Form (IPAQ-SF)
Cardiorespiratory fitness | Baseline
  Pulmonary maximal oxygen uptake (VO2max) is determined during an incremental exercise test to exhaustion

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Fiorenza, Ph.D., Principal Investigator — Rigshospitalet, Denmark; John Vissing, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeFronzo RA, Ferrannini E. Insulin resistance. A multifaceted syndrome responsible for NIDDM, obesity, hypertension, dyslipidemia, and atherosclerotic cardiovascular disease. Diabetes Care. 1991 Mar;14(3):173-94. doi: 10.2337/diacare.14.3.173. PMID 2044434
- [Background] DeFronzo RA, Simonson D, Ferrannini E. Hepatic and peripheral insulin resistance: a common feature of type 2 (non-insulin-dependent) and type 1 (insulin-dependent) diabetes mellitus. Diabetologia. 1982 Oct;23(4):313-9. doi: 10.1007/BF00253736. PMID 6754515
- [Background] DeFronzo RA, Gunnarsson R, Bjorkman O, Olsson M, Wahren J. Effects of insulin on peripheral and splanchnic glucose metabolism in noninsulin-dependent (type II) diabetes mellitus. J Clin Invest. 1985 Jul;76(1):149-55. doi: 10.1172/JCI111938. PMID 3894418
- [Background] Diaz-Vegas A, Sanchez-Aguilera P, Krycer JR, Morales PE, Monsalves-Alvarez M, Cifuentes M, Rothermel BA, Lavandero S. Is Mitochondrial Dysfunction a Common Root of Noncommunicable Chronic Diseases? Endocr Rev. 2020 Jun 1;41(3):bnaa005. doi: 10.1210/endrev/bnaa005. PMID 32179913
- [Background] Hesselink MK, Schrauwen-Hinderling V, Schrauwen P. Skeletal muscle mitochondria as a target to prevent or treat type 2 diabetes mellitus. Nat Rev Endocrinol. 2016 Nov;12(11):633-645. doi: 10.1038/nrendo.2016.104. Epub 2016 Jul 22. PMID 27448057
- [Background] Parish R, Petersen KF. Mitochondrial dysfunction and type 2 diabetes. Curr Diab Rep. 2005 Jun;5(3):177-83. doi: 10.1007/s11892-005-0006-3. PMID 15929863
- [Background] Zabielski P, Lanza IR, Gopala S, Heppelmann CJ, Bergen HR 3rd, Dasari S, Nair KS. Altered Skeletal Muscle Mitochondrial Proteome As the Basis of Disruption of Mitochondrial Function in Diabetic Mice. Diabetes. 2016 Mar;65(3):561-73. doi: 10.2337/db15-0823. Epub 2015 Dec 30. PMID 26718503
- [Background] Petersen MC, Shulman GI. Mechanisms of Insulin Action and Insulin Resistance. Physiol Rev. 2018 Oct 1;98(4):2133-2223. doi: 10.1152/physrev.00063.2017. PMID 30067154
- [Background] O'Rahilly S. "Treasure Your Exceptions"-Studying Human Extreme Phenotypes to Illuminate Metabolic Health and Disease: The 2019 Banting Medal for Scientific Achievement Lecture. Diabetes. 2021 Jan;70(1):29-38. doi: 10.2337/dbi19-0037. PMID 33355307
- [Background] Saleheen D, Natarajan P, Armean IM, Zhao W, Rasheed A, Khetarpal SA, Won HH, Karczewski KJ, O'Donnell-Luria AH, Samocha KE, Weisburd B, Gupta N, Zaidi M, Samuel M, Imran A, Abbas S, Majeed F, Ishaq M, Akhtar S, Trindade K, Mucksavage M, Qamar N, Zaman KS, Yaqoob Z, Saghir T, Rizvi SNH, Memon A, Hayyat Mallick N, Ishaq M, Rasheed SZ, Memon FU, Mahmood K, Ahmed N, Do R, Krauss RM, MacArthur DG, Gabriel S, Lander ES, Daly MJ, Frossard P, Danesh J, Rader DJ, Kathiresan S. Human knockouts and phenotypic analysis in a cohort with a high rate of consanguinity. Nature. 2017 Apr 12;544(7649):235-239. doi: 10.1038/nature22034. PMID 28406212
- [Background] DiMauro S. Mitochondrial myopathies. Curr Opin Rheumatol. 2006 Nov;18(6):636-41. doi: 10.1097/01.bor.0000245729.17759.f2. PMID 17053512
- [Background] Gorman GS, Schaefer AM, Ng Y, Gomez N, Blakely EL, Alston CL, Feeney C, Horvath R, Yu-Wai-Man P, Chinnery PF, Taylor RW, Turnbull DM, McFarland R. Prevalence of nuclear and mitochondrial DNA mutations related to adult mitochondrial disease. Ann Neurol. 2015 May;77(5):753-9. doi: 10.1002/ana.24362. Epub 2015 Mar 28. PMID 25652200
- [Background] Elliott HR, Samuels DC, Eden JA, Relton CL, Chinnery PF. Pathogenic mitochondrial DNA mutations are common in the general population. Am J Hum Genet. 2008 Aug;83(2):254-60. doi: 10.1016/j.ajhg.2008.07.004. PMID 18674747
- [Background] Frederiksen AL, Jeppesen TD, Vissing J, Schwartz M, Kyvik KO, Schmitz O, Poulsen PL, Andersen PH. High prevalence of impaired glucose homeostasis and myopathy in asymptomatic and oligosymptomatic 3243A>G mitochondrial DNA mutation-positive subjects. J Clin Endocrinol Metab. 2009 Aug;94(8):2872-9. doi: 10.1210/jc.2009-0235. Epub 2009 May 26. PMID 19470628
- [Background] Lindroos MM, Majamaa K, Tura A, Mari A, Kalliokoski KK, Taittonen MT, Iozzo P, Nuutila P. m.3243A>G mutation in mitochondrial DNA leads to decreased insulin sensitivity in skeletal muscle and to progressive beta-cell dysfunction. Diabetes. 2009 Mar;58(3):543-9. doi: 10.2337/db08-0981. Epub 2008 Dec 10. PMID 19073775